CLINICAL TRIAL: NCT02089620
Title: Calcium Supplements Versus Oral Contraceptive Pills Containing Drospirenone in Treating Mild to Moderate Premenstrual Syndrome: A Double Blind Randomized Placebo Controlled Trial
Brief Title: Comparison Between Oral Contraceptive Pills and Calcium Supplements in Treatment of Premenstrual Syndrome
Acronym: PMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Nesreen Abdel Fattah Abdullah Shehata, Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Beni-Suef 1
Record Dates: First submitted 2014-03-02; First posted 2014-03-18 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; Oral contraceptive pills; Calcium Supplements
MeSH Terms: conditions — Premenstrual Syndrome | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yasmin (Active Comparator): Yasmin is an oral contraceptive pill containing (Disperinone 3mg+Ethinylestradiol 0.3mg) will be administered once daily orally by the woman from day 2 of the cycle for 21 days each month for 3 months in addition to a daily placebo.
  Interventions: Drug: Yasmin; Drug: Placebo 1
- Calver (Active Comparator): Calver is a calcium supplement drug containing (ca 1000mg+vit D400 I.U) given to the woman continuously for 3 months in addition to placebo for 21 days
  Interventions: Dietary Supplement: Calver; Drug: Placebo 2
- Placebo (Placebo Comparator): A daily oral placebo will be given to the patients daily for 3 months in addition to a placebo similar to COC for 21 days
  Interventions: Drug: Placebo 1; Drug: Placebo 2

INTERVENTIONS:
Drug: Yasmin — will be used every 21 days for three months by the patient
  Other Names: OCP
  Arms: Yasmin
Dietary Supplement: Calver — Calver will be given daily for 3 months
  Other Names: Calcium supplement
  Arms: Calver
Drug: Placebo 1 — Patients will receive a daily placebo similar in size and structure to calvar.
  Arms: Placebo; Yasmin
Drug: Placebo 2 — Women will receive an oral placebo similar to COC for 21 days starting from the 3rd day of menstruation
  Arms: Calver; Placebo

SUMMARY:
Premenstrual syndrome represents a group of problems affecting most of women in reproductive age. These problems include emotional and physical symptoms. In this study the efficacy of oral contraceptive pills and calcium supplements in relieving these symptoms will be assessed .

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is deﬁned as the recurrence of psychological and physical symptoms in the luteal phase, which remit in the follicular phase of the menstrual cycle [1].PMS will be prospectively diagnosed using the Royal college of Obstetricians and Gynecologists (RCOG) recommended daily record of severity of problems (DRSP) . Women will be asked to fill the diary for 2 months, only women with 30% increase in the DRSP score in the week before menses in both months will be diagnosed as having PMS.

Women with PMS will be invited to participate in the study.The invitation will include a clear full explanation of the study and patients will provide written consents. All patients consenting to participate will be included in the trial.

Yasmin, Calver and Placebo will be enclosed in sequentially numbered similar bottles which will be numbered using a computer generated random table. Women will be asked to choose a sealed envelope, each envelope will contain the number allocated to the jar and special instructions on how to use the medication. Yasmin will be taken once daily for 21 days starting from the 2nd day of menstruation, Calver and placebo will be taken continuously. Neither the patients nor the physician will be aware of the drug used. Patients will be categorized in 3 groups: group1 who will receive Yasmin cyclically for 3 months (Yasmin, schering, cairo, Egypt) and daily oral placebo, group 2 who will receive Calver continuously for 3 months (Calver, Marcryl/Vertex, Cairo Egypt) and oral placebo for 21 days, group 3 who will receive a daily placebo and a placebo similar to COC for 21 days and will act as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed by prospective dairy to have PMS
* Consenting to be included in the study
* Age 18-40 years

Exclusion Criteria:

* Medical disorders as hypertension or diabetes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Improvement of premenstrual symptoms. | 3 months after starting treatment.
  Improvement of symptoms will be assessed by comparing the pre-treatment recorded DRSP with that recorded 3 months after starting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen A Shehata, Lecturer, Principal Investigator — Beni-Suef University; Abdelgany M Hassan, Lecturer, Study Chair — Cairo University
Locations (1):
- Beni-Suef University, Banī Suwayf, Egypt

REFERENCES:
- [Background] Endicott J, Nee J, Harrison W. Daily Record of Severity of Problems (DRSP): reliability and validity. Arch Womens Ment Health. 2006 Jan;9(1):41-9. doi: 10.1007/s00737-005-0103-y. Epub 2005 Sep 20. PMID 16172836
- [Background] Wyatt K, Dimmock P, Jones P, Obhrai M, O'Brien S. Efficacy of progesterone and progestogens in management of premenstrual syndrome: systematic review. BMJ. 2001 Oct 6;323(7316):776-80. doi: 10.1136/bmj.323.7316.776. PMID 11588078
- [Derived] Shehata NAA. RETRACTED: Calcium versus oral contraceptive pills containing drospirenone for the treatment of mild to moderate premenstrual syndrome: a double blind randomized placebo controlled trial. Eur J Obstet Gynecol Reprod Biol. 2016 Mar;198:100-104. doi: 10.1016/j.ejogrb.2016.01.015. Epub 2016 Jan 13. PMID 26808666 (Retraction: PMID 31455589 Eur J Obstet Gynecol Reprod Biol. 2019 Sep;240:387)